CLINICAL TRIAL: NCT06905119
Title: Digital Transformation of Continuity of Care for Peripherally Inserted Central Catheters: SpadCare Experience
Acronym: SpadCare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Universidad Pública de Navarra (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38_NAV2
Record Dates: First submitted 2025-02-19; First posted 2025-04-01 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Infusions, Intravenous; Administration, Intravenous; Home Infusion Therapy; Parenteral Nutrition, Home; Central Venous Catheters; Catheterization, Central Venous; Catheterization, Peripheral; Vascular Access Devices; Patient Education as Topic; Patient Participation; User-Computer Interface; Smartphone; Mobile Applications; Computers, Handheld; Digital Health; Nursing; Care Givers; Delivery of Health Care; Home Nursing; Self Administration; Adverse Effects; Catheter-Related Infections; Telemedicine
Keywords: Catheterization, Peripheral; Vascular Access Devices; Patient Education as Topic; Telemedicine; Mobile Applications
MeSH Terms: conditions — Hyperphagia; Patient Participation; Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smart phone APP (Experimental): Patients who agree to participate in the study, once the PICC is placed, download the app to their personal Smartphone or that of a family member. The app contains all the information about the catheter, including the insertion date, gauge, number of lumens, batch number, and more. The weekly catheter care is performed at home, at the health center, or in the hospital and can be performed by nursing professionals or properly trained family members or caregivers of the patient. The patient reports any incidents that may occur each week. If an incident occurs, the responsible professional contacts the patient by phone and, if necessary, makes an appointment for an in-person consultation to review the catheter. The patient records the care performed in the app and a reminder is automatically recorded in the phone calendar. The app has documentation prepared by expert personnel along with video procedures for the care, and the "step-by-step" feature that allows the care to be performed.
  Interventions: Other: Digital Transformation of Continuity of Care for Peripherally Inserted Central Catheters
- Control arm (No Intervention): Usual care description: Patients in the intervention group only have information about their catheter (placement date, catheter reference and batch) on a paper card; they do not have documentary or audiovisual resources. The treatment is carried out exclusively by nursing professionals at the hospital or health centre, and the latter are the ones who contact the hospital professionals who placed it in the event of an incident. The professionals who inserted the catheter are aware of the information about the catheter removal and whether there has been any significant complication when reviewing the catheters they have inserted at the end of the year, and are not aware of the incidents until the annual review. The under-registration in computer applications means that information on a high number of inserted catheters is not available.

INTERVENTIONS:
Other: Digital Transformation of Continuity of Care for Peripherally Inserted Central Catheters — The application is offered to all patients at the time of PICC placement. If they accept, they go to the intervention group. If they do not accept, they go to the control group.
  Other Names: SpadCare Experience
  Arms: Smart phone APP

SUMMARY:
The study focuses on patients who require outpatient infusion of therapy ("Infusions, Intravenous"[Mesh]) "Administration, Intravenous"[Mesh] ("Home Infusion Therapy"[Mesh]) "Parenteral Nutrition, Home"[Mesh] via a peripherally inserted central catheter (PICC) ("Central Venous Catheters"[MeSH] "Catheterization, Central Venous"[MeSH] "Catheterization, Peripheral" [MeSH] "Vascular Access Devices"[Mesh] )

DETAILED DESCRIPTION:
The patients, who receive training ("Patient Education as Topic"[Mesh] "patient participation"[MeSH Terms] ) via an app on their personal mobile phone ("User-Computer Interface"[Mesh] "Smartphone"[MeSH] "Mobile Applications"[MeSH] "Computers, Handheld"[Mesh] "Digital Health"[Mesh] are able to perform specialized care ("Nursing"[Mesh]) Care"[MeSH] "Delivery of Health Care"[Mesh:NoExp] "Home Nursing"[MeSH] "Self Administration"[Mesh] to reduce complications ("adverse effects"[MeSH Subheading] "Catheter-Related Infections"[Mesh] ) so that they are monitored in real time by those responsible for the catheter. ("Telemedicine"[Mesh]

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years.
* Sign the informed consent form.
* Have a Smartphone and accept the use of the APP.
* Patient with a PICC inserted by the Infusion and Vascular Access Team of the University Hospital of Navarra and with a planned use of at least one month.

Exclusion Criteria:

* Patients with limitations in the use of digital resources or lack of Smartphone.
* Patients who do not want to install the APP on their Smartphone
* Patients who do not authorize access to their Computerized Medical Record (HCI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
1. Patients who use computerized applications are more involved in their care and have fewer complications with the PICC | At the end of intervention: Time from PICC placement to removal.
  Number of phlebitis episodes
1. Patients who use computerized applications are more involved in their care and have fewer complications with the PICC. | At the end of intervention: Time from PICC placement to removal.
  Number of episodes of catheter removal by reason for removal: pain
1. Patients who use computerized applications are more involved in their care and have fewer complications with the PICC. | At the end of intervention: Time from PICC placement to removal.
  Number of infection episodes
1. Patients who use computerized applications are more involved in their care and have fewer complications with the PICC. | At the end of the intervention: Time from PICC placement to removal.
  Number of episodes of withdrawal reason due to accidental exit
1. Patients who use computerized applications are more involved in their care and have fewer complications with the PICC. | At the end of intervention: Time from PICC placement to removal.
  Number of episodes of skin lesions
1. Patients who use computerized applications are more involved in their care and have fewer complications with the PICC. | At the end of intervention: Time from PICC placement to removal.
  Number of thrombosis episodes
1. Patients who use computerized applications are more involved in their care and have fewer complications with the PICC. | At the end of intervention: Time from PICC placement to removal.
  Number of episodes of catheter breakage as a reason for removal

SECONDARY OUTCOMES:
Patient experience | At the end of using the application: Time from PICC placement to removal.
  Patient satisfaction with the use of the app, through the questionnaire CSUQ: Computer System Usability Questionnaire. The CSUQ scale, or System Usability Satisfaction Questionnaire, is a tool used to assess user satisfaction with a specific system. It is a Likert-type measurement scale, where participants evaluate their level of satisfaction with various aspects of a system, generally on a scale ranging from 1 (totally disagree) to 7 (totally agree).
Patient experience | At the end of using the application: Time from PICC placement to removal.
  Patient satisfaction with the use of the app, through the questionnaire eHEALS. The eHealth Literacy Scale (eHEALS) is a tool that measures eHealth literacy by assessing individuals' subjective perception of their skills and knowledge in using online health resources. The questionnaire consists of eight questions that are answered on a Likert scale, where scores range from 1 (Strongly disagree) to 5 (Strongly agree).
Patient Satisfaction | At the end of using the application: Time from PICC placement to removal.
  Overall satisfaction questionnaire with SpadCare, generated by the research team.
  SpadCare Questionnaire: 1 the worst value to 10 the best value How would you rate the SpadCare application you have just tested? From 1 to 10, where 1 means 'very dissatisfied' and 10 means 'very satisfied' How likely are you to recommend it to other patients?

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No